CLINICAL TRIAL: NCT00196339
Title: A Dose-ranging Clinical Trial to Study the Efficacy and Safety of DR-2031 for the Treatment of Hot Flashes Following Surgical or Medical Castration of Prostate Cancer Patients
Brief Title: A Clinical Trial to Study DR-2031 for the Treatment of Hot Flashes in Prostate Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duramed Research (Industry)
Responsible Party: Sponsor
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DR-PCA-201
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2016-07-22 (Estimated); Status verified 2016-07

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; hot flashes; hot flushes; vasomotor symptoms
MeSH Terms: conditions — Prostatic Neoplasms; Hot Flashes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Cyproterone acetate 5 mg ( DR-2031) (Experimental): 1 tablet daily
  Interventions: Drug: Cyproterone acetate 5
- Cyproterone acetate 15 mg ( DR-2031) (Experimental): 1 tablet daily
  Interventions: Drug: Cyproterone acetate 15
- Cyproterone acetate 25 mg ( DR-2031) (Experimental): 1 tablet daily
  Interventions: Drug: Cyproterone acetate 25
- Placebo (Placebo Comparator): 1 tablet daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cyproterone acetate 5 — Cyproterone acetate 5 mg
  Other Names: DR-2031
  Arms: Cyproterone acetate 5 mg ( DR-2031)
Drug: Placebo — Matching placebo
  Arms: Placebo
Drug: Cyproterone acetate 15 — Cyproterone acetate 15 mg
  Other Names: DR-2031
  Arms: Cyproterone acetate 15 mg ( DR-2031)
Drug: Cyproterone acetate 25 — Cyproterone acetate 25 mg
  Other Names: DR-2031
  Arms: Cyproterone acetate 25 mg ( DR-2031)

SUMMARY:
This is a study to compare the efficacy and safety of 3 doses of DR-2031 to placebo when used as "add-on" therapy for prostate cancer patients with hot flashes following surgical or medical castration. All prostate cancer therapy must be stable for at least 45 days before entering the study and must remain stable throughout this 12-week study. Patients will maintain a daily paper diary to record the frequency and severity of hot flashes during the treatment period.

DETAILED DESCRIPTION:
This is a study to compare the efficacy and safety of 3 doses of DR-2031 to placebo when used as "add-on" therapy for prostate cancer in patients with mild to moderate vasomotor symptoms (hot flashes) following surgical or medical castration. All prostate cancer therapy must be stable for at least 45 days before entering the study and must remain stable throughout this 12-week study. To be eligible for this study prostate cancer patients must have undergone bilateral orchiectomy or medical castration utilizing LHRH analogues (LHRH agonists or LHRH antagonists) with or without additional antiandrogen therapy. Patients must have at least 21 moderate to severe hot flashes weekly.

Patients will maintain a daily paper diary to record the frequency and severity of hot flashes during the treatment period. In addition, a brief physical evaluation will be done, diaries will be reviewed and any adverse events will be recorded at each follow-up evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer patients who have undergone chemical or surgical castration
* History of hot flashes for at least 30 days
* Stable prostate cancer therapy for at least 45 days

Exclusion Criteria:

* Uncontrolled diabetes or severe COPD
* History of thromboembolic disease
* Liver or kidney dysfunction
* History or presence of cancer other than prostate cancer within the last 5 years
* Surgery within the last 3 months

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315 (Actual)
Dates: Start 2005-06; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy in reducing the frequency and severity of moderate to severe hot flashes | Throughout study
To evaluate the safety compared to placebo | Throughout study
Identify the lowest effective dose. | End of study

SECONDARY OUTCOMES:
To compare the efficacy in reducing the severity of all hot flashes | Throughout study
To compare the efficacy in elimination of all hot flashes | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Duramed Protocol Chair, Study Chair — Duramed Research, Inc.
Locations (109):
- United States (91):
  - Duramed Investigational Site, Birmingham, Alabama
  - Duramed Investigational Site, Homewood, Alabama
  - Duramed Investigational Site, Huntsville, Alabama
  - Duramed Investigational Site, Phoenix, Arizona
  - Duramed Investigational Site, Tucson, Arizona
  - Duramed Investigational Site, Little Rock, Arkansas
  - Duramed Investigational Site, Anaheim, California
  - Duramed Investigational Site, Fresno, California
  - Duramed Investigational Site, La Mesa, California
  - Duramed Investigational Site, Laguna Hills, California
  - Duramed Investigational Site, Laguna Woods, California
  - Duramed Investigational Site, Long Beach, California
  - Duramed Investigational Site, Los Angeles, California
  - Duramed Investigational Site, San Bernardino, California
  - Duramed Investigational Site, San Diego, California
  - Duramed Investigational Site, Torrance, California
  - Duramed Investigational Site, Denver, Colorado
  - Duramed Investigational Site, Wheat Ridge, Colorado
  - Duramed Investigational Site, Middlebury, Connecticut
  - Duramed Investigational Site, New Britain, Connecticut
  - Duramed Investigational Site, Trumbull, Connecticut
  - Duramed Investigational Site, Waterbury, Connecticut
  - Duramed Investigational Site, Washington D.C., District of Columbia
  - Duramed Investigational Site, Aventura, Florida
  - Duramed Investigational Site, Daytona Beach, Florida
  - Duramed Investigational Site, New Port Richey, Florida
  - Duramed Investigational Site, Ocala, Florida
  - Duramed Investiational Site, Ocala, Florida
  - Duramed Investigational Site, Plantation, Florida
  - Duramed Investigational Site, Sarasota, Florida
  - Duramed Investigational Site, Spring Hill, Florida
  - Duramed Investigational Site, St. Petersburg, Florida
  - Duramed Investigational site, Atlanta, Georgia
  - Duramed Investigational Site, Coeur d'Alene, Idaho
  - Duramed Investigational Site, Berwyn, Illinois
  - Duramed Investigational Site, Chicago, Illinois
  - Duramed Investigational Site, Kankakee, Illinois
  - Duramed Investigational Site, Peoria, Illinois
  - Duramed Investigational Site, Greenwood, Indiana
  - Duramed Investigational Site, Jeffersonville, Indiana
  - Duramed Investigational Site, Des Moines, Iowa
  - Duramed Investigational Site, Overland Park, Kansas
  - Duramed Investigational Site, New Orleans, Louisiana
  - Duramed Investigational Site, Shreveport, Louisiana
  - Duramed Investigational Site, Greenbelt, Maryland
  - Duramed Investigational Site, Newton, Massachusetts
  - Duramed Investigational Site, Watertown, Massachusetts
  - Duramed Investigational Site, Saint Joseph, Michigan
  - Duramed Investigational Site, Sartell, Minnesota
  - Duramed Investigational Site, Jackson, Mississippi
  - Duramed Investigational Site, St Louis, Missouri
  - Duramed Investigational Site, Las Vegas, Nevada
  - Duramed Investigational Site, Brick, New Jersey
  - Duramed Investigational Site, Edison, New Jersey
  - Duramed Investigational Site, Lawrenceville, New Jersey
  - Duramed Investigational Site, Albany, New York
  - Duramed Investigational Site, Bay Shore, New York
  - Duramed Investigational Site, Elmont, New York
  - Duramed Investigational site, Garden City, New York
  - Duramed Investigational Site, New York, New York
  - Duramed Investigational Site, Poughkeepsie, New York
  - Duramed Investigational Site, Staten Island, New York
  - Duramed Investigational Site, Williamsville, New York
  - Duramed Investigational Site, Asheboro, North Carolina
  - Duramed Investigational Site, Concord, North Carolina
  - Duramed Investigational Site, Raleigh, North Carolina
  - Duramed Investigational Site, Fargo, North Dakota
  - Duramed Investigational Site, Canfield, Ohio
  - Duramed Investigational Site, Canton, Ohio
  - Duramed Investigational Site, Cincinnati, Ohio
  - Duramed Investigational Site, Bethany, Oklahoma
  - Duramed Investigational Site, Oklahoma City, Oklahoma
  - Duramed Investigational Site, Allentown, Pennsylvania
  - Duramed Investigational Site, Bala-Cynwyd, Pennsylvania
  - Duramed Investigational Site, Lancaster, Pennsylvania
  - Duramed Investigational Site, Philadelphia, Pennsylvania
  - Duramed Investigational Site, Pittsburgh, Pennsylvania
  - Duramed Investigational Site, Sellersville, Pennsylvania
  - Duramed Investigational Site, State College, Pennsylvania
  - Duramed Investigational Site, Providence, Rhode Island
  - Duramed Investigational Site, Charleston, South Carolina
  - Duramed Investigational Site, Knoxville, Tennessee
  - Duramed Investigational Site, Austin, Texas
  - Duramed Investigational Site, Dallas, Texas
  - Duramed Investigational Site, Houston, Texas
  - Duramed Investigational Site, San Antonio, Texas
  - Duramed Investigational Site, Salt Lake City, Utah
  - Duramed Investigational Site, Richmond, Virginia
  - Duramed Investigational Site, Seattle, Washington
  - Duramed Investigational Site, Tacoma, Washington
  - Duramed Investigational Site, Milwaukee, Wisconsin
- Canada (18):
  - Duramed Investigational Site, Kelowna, British Columbia
  - Duramed Investigational Site, Surrey, British Columbia
  - Duramed Investigational Site, Vancouver, British Columbia
  - Duramed Investigational Site, Victoria, British Columbia
  - Duramed Investigational Site, Saint John, New Brunswick
  - Duramed Investigational Site, Kentville, Nova Scotia
  - Duramed Investigational Site, Barrie, Ontario
  - Duramed Investigational Site, Brantford, Ontario
  - Duramed Investigational Site, Greater Sudbury, Ontario
  - Duramed Investigational Site, Guelph, Ontario
  - Duramed Investigational Site, Markham, Ontario
  - Duramed Investigational Site, North Bay, Ontario
  - Duramed Investigational Site, Oakville, Ontario
  - Duramed Investigational Site, Oshawa, Ontario
  - Duramed Investigational Site, Ottawa, Ontario
  - Duramed Investigational Site, Toronto, Ontario
  - Duramed Investigational Site, Mirabel, Quebec
  - Duramed Investigational Site, Pointe-Claire, Quebec

REFERENCES:
- See also: MedLine Plus - Prostate Cancer — http://www.nlm.nih.gov/medlineplus/prostatecancer.html